CLINICAL TRIAL: NCT01863277
Title: A Double Blind, Placebo Controlled Study to Evaluate the Efficacy of Melatonin in Acute Ischemic Stroke.
Brief Title: Safety Study of Melatonin in Stroke Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Yair Lampl, Prof. Yair Lampl, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0130-12
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-04

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin (Active Comparator): Melatonin 14mg/daily given over 14 days
  Interventions: Drug: Melatonin
- sugar pill (Placebo Comparator): sugar pill given over 14 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Melatonin
  Arms: Melatonin
Drug: placebo
  Arms: sugar pill

SUMMARY:
The purpose of the study is to evaluate the effect of Melatonin (in a dosage of 14mg daily) for a better clinical outcome in the period three days post stroke.

DETAILED DESCRIPTION:
Stroke is the third most common cause of stroke. The cascade of event is separated into hyperacute,,acute,sub-acute and chronic. In the acute, sub acute state there are mechanisms of inflammation apoptotic death and effect of free radicals. Melatonin was proved to effect these mechanisms and to have a favourable effect in different diseases. The aim of the study is to prove That the use of Melatonin in a higher dosage may have a anti-destructive effect in stoke.

ELIGIBILITY:
Inclusion Criteria:

* within 72hours of ischemic stroke
* age 18-80
* both gender
* ability to sign consent form

Exclusion Criteria:

* intra-cerebral bleeding
* tumour of brain
* multiple sclerosis
* s/p craniotomy
* known allergy to melatonin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Improvement of at least one point on the MRS score | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- E. Wolfson Medical Center, Holon, Israel